CLINICAL TRIAL: NCT04183361
Title: Correlation of Auditory Evoked Brainstem Response Characteristics and Salivary Cortisone Concentration in Noise-exposed Workers
Brief Title: ABR Characteristics and Salivary Cortisone Concentration in Noise-exposed Workers
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Andro Košec, MD, PhD, Consultant Otorhinolaryngologist and Head and Neck Surgeon, University Hospital Sestre Milosrdnice
Other Study IDs: EP-ABR01
Record Dates: First submitted 2019-11-27; First posted 2019-12-03 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Sensorineural Hearing Loss; Noise Induced Hearing Loss; Auditory Nerve; Lesion
Keywords: noise; sensorineural hearing loss; ABR; cortisole; salivary
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Noise-Induced; Vestibulocochlear Nerve Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Three saliva samples at the workplace immediately after the morning shift. The first saliva sample was given 3 days (Tuesday) before arrival at the research place, the second sample 2 days (Wednesday) before arrival, and the third sample 1 day (Thursday) before arrival at the research site. Coded saliva samples in laboratory by using High Performance Liquid Chromatography (HPLC) at the Translational Medicine Division of the Srebrnjak Children's Hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with noise exposure and salivary cortisone: 1. male and female
  2. ages 19-35
  3. exposure to noise level ≥ 85 dB (A) per week at the workplace
  4. work in noise from 1 to 16 years
  5. workplace not involving exposure to carbon disulfide or a mixture of organic solvents that have toxic effects on the ear (toluene, xylene and styrene)
  6. unilaterally or bilaterally normal otoscopic findings
  7. unilaterally or bilaterally tympanogram: peak pressure value ± 50 daPa at 226 Hz with eardrum mobility of 0.3 to 1.3 mL
  Interventions: Diagnostic Test: ABR and salivary cortisone testing
- Patients without noise exposure and salivary cortisone: 1. male and female
  2. ages 19-35
  3. no exposure to noise level ≥ 85 dB (A) per week at the workplace
  4. work in noise from 1 to 16 years
  5. workplace not involving exposure to carbon disulfide or a mixture of organic solvents that have toxic effects on the ear (toluene, xylene and styrene)
  6. unilaterally or bilaterally normal otoscopic findings
  7. unilaterally or bilaterally tympanogram: peak pressure value ± 50 daPa at 226 Hz with eardrum mobility of 0.3 to 1.3 mL
  Interventions: Diagnostic Test: ABR and salivary cortisone testing

INTERVENTIONS:
Diagnostic Test: ABR and salivary cortisone testing — Three saliva samples at the workplace will be collected immediately after the morning shift. The first saliva sample was given 3 days (Tuesday) before arrival at the research place, the second sample 2 days (Wednesday) before arrival, and the third sample 1 day (Thursday) before arrival at the research site. One hour before saliva sampling, a respondent should not brush his/her teeth nor eat nor drink. Fifteen minutes prior to sample administration, the subject should rinse his/her mouth with a cold water. Samples will be analyzed using High Performance Liquid Chromatography (HPLC) at the Translational Medicine Division of the Srebrnjak Children's Hospital.
  2. Collaboration in the process of assessing hearing health at the research place. The assessment includes: otoscopy, tympanometry and audiometry. Subjects will be tested for auditory evoked brainstem response in only one ear, with a more regular hearing threshold.

SUMMARY:
The aim of the research:

Investigate the association of auditory evoked brainstem response characteristics with salivary cortisone concentrations in noise-exposed workers.

Purpose of the research:

1. Investigate the magnitude of the amplitudes and latencies of auditory brainstem responses.
2. Investigate the concentration of cortisone in saliva.
3. To investigate the correlation of the characteristics of auditory evoked brainstem potentials with the age of the subjects or the length of work in noise.
4. Investigate the association of salivary cortisone concentration with subjects' age or length of work in noise.
5. Investigate the prevalence of mild, moderate and severe hearing impairment in the 19-35 age group.
6. Investigate the relationship of hearing threshold shift with the age of the subjects or the length of work in noise.
7. To investigate the difference in the characteristics of auditory evoked brainstem potentials and the difference in salivary cortisone concentration between subjects with a bilaterally normal hearing threshold (≤25 dB) at high frequencies and subjects with unilaterally or bilaterally increased hearing threshold (> 25 dB) at high frequencies .
8. Investigate the perceived stress and psychosocial risk factors in the workplace and their relationship to salivary cortisone concentrations.

Research Hypothesis:

There is an association between the characteristics of auditory evoked brainstem response and salivary cortisone concentrations in noise-exposed workers.

Research participants

Inclusion criteria:

1. male and female
2. ages 19-35
3. exposure to noise level ≥ 85 dB (A) per week at the workplace
4. work in noise from 1 to 16 years
5. workplace not involving exposure to carbon disulfide or a mixture of organic solvents that have toxic effects on the ear (toluene, xylene and styrene)
6. unilaterally or bilaterally normal otoscopic findings
7. unilaterally or bilaterally tympanogram: peak pressure value ± 50 daPa at 226 Hz with eardrum mobility of 0.3 to 1.3 mL

Exclusion criteria:

1. information about an earlier sudden hearing loss
2. information on chronic middle ear inflammation
3. information on ear surgery (except placement of ventilation tubes in the eardrum)
4. information on dizziness associated with hearing loss and noise
5. information on insomnia
6. current use of oral corticosteroids
7. bilaterally found air-bone gap greater than 15 dB

DETAILED DESCRIPTION:
The research is cross-sectional. The expected duration of the survey is at least 18 months. Assuming that the characteristics of the auditory evoked brainstem potentials are correlated with salivary cortisone concentration with a correlation coefficient of 0.4, a test power of 80% and a significance level of α = 0.05, at least 46 subjects should be included in the study. Test power analysis was performed using MedCalc Statistical Software, version 19.1 (MedCalc Software bv, Ostend, Belgium; https://www.medcalc.org; 2019). According to the data distribution (Kolmogorov-Smirnov test), appropriate parametric and / or non-parametric statistical tests will be applied in accordance with the obtained results. The data will be presented in tables and graphs. Numerical variables will be represented using the range, arithmetic mean and standard deviation, respectively, the median and the interquartile range, in cases of distribution that does not follow the normal distribution. The categorical variables will be presented using absolute frequencies and their respective proportions. Differences in the values of the numerical variables between the test groups with a defined hearing threshold will be analyzed by parametric Student's t-test for independent samples, and non-parametric Mann-Whitney U test for independent samples. Differences in categorical variables between the examined groups will be analyzed by chi-square test or Fisher's exact test in cases where the number of subjects in each group is less than 5. The corresponding correlation coefficients (Pearson's or Spearman's) between individual clinical variables will be calculated. An appropriate regression model for the prediction of belonging to a group with a defined hearing threshold shift will be made, which will include those that have a significance level of P≤0.20 in the previous statistical analyzes. In the above tests, significant P values will be considered to be less than 0.05. The statistical analysis of data will use IBM SPSS Statistics licensed software version 25.0.

Material:

1. Audiometer Audiometer AC40
2. DD45 audiometric headphones
3. Interacoustics AZ26 tympanometer
4. Equipment for testing auditory evoked brainstem potentials: ABR Interacoustics Eclipse, EPA Preamplifier, 3M E-A-RTONE Insert Earphone ABR
5. Cortisol-Salivette Cotton Salad Carrier
6. High Performance Liquid Chromatography (HPLC)
7. validated questionnaire in the Croatian language - assessment of psychosocial risk factors in the HSE workplace 8th validated questionnaire in Croatian - The scale of stress experienced

Research plan:

An employer finds workers who meet points 1-5 of study inclusion criteria. A head of the research checks their medical history and includes them in the study if they do not meet any of first six exclusion criteria. A head of the research orally informs these workers at the meeting and helps them to understand and sign a written informed consent for participation in the research. Each of them receive an information about the date of arrival at the place of research and also a unique password that encodes saliva samples, completed questionnaires and electronic and printed findings derived from the assessment of hearing health. The research leader, research mentors, and occupational safety manager, who is responsible for supervising the sampling and storage of saliva samples in the refrigerator at +4 ℃ in the workplace, know the password and associated name.

A participant is expected to:

1. Give three saliva samples at the workplace immediately after the morning shift. The first saliva sample was given 3 days (Tuesday) before arrival at the research place, the second sample 2 days (Wednesday) before arrival, and the third sample 1 day (Thursday) before arrival at the research site. One hour before saliva sampling, a respondent should not brush his/her teeth nor eat nor drink. Fifteen minutes prior to sample administration, the subject should rinse his/her mouth with a cold water. Then head of the research analyses coded saliva samples in laboratory by using High Performance Liquid Chromatography (HPLC) at the Translational Medicine Division of the Srebrnjak Children's Hospital. After processing and preparing each of the saliva samples for HPLC, the native sample no longer exists. After the analytes will be detected in the isolate, all the material will be completely eliminated as infectious waste.
2. Collaboration in the process of assessing hearing health at the research place. The assessment includes: otoscopy, tympanometry and audiometry. Subjects who do not meet point 6 and 7 of the inclusion criteria or who meet point 7 of the exclusion criteria will not be tested for auditory evoked brainstem response. Other subjects will be tested for auditory evoked brainstem response in only one ear, with a more regular hearing threshold.
3. Self-assessment of perceived stress and psychosocial risk factors in the workplace by completing a questionnaire at the research site.

A researcher conducting this research and the research participants will not receive a financial fee for their participation.

Expected scientific contribution of the research:

Quantification of the association of auditory evoked brainstem response characteristics with salivary cortisone concentrations among workers exposed to noise.

Possible risks of participating in the research:

This research involves no risk other than the usual daily risk.

ELIGIBILITY:
Inclusion Criteria:

1. male and female
2. ages 19-35
3. exposure to noise level ≥ 85 dB (A) per week at the workplace
4. work in noise from 1 to 16 years
5. workplace not involving exposure to carbon disulfide or a mixture of organic solvents that have toxic effects on the ear (toluene, xylene and styrene)
6. unilaterally or bilaterally normal otoscopic findings
7. unilaterally or bilaterally tympanogram: peak pressure value ± 50 daPa at 226 Hz with eardrum mobility of 0.3 to 1.3 mL

Exclusion Criteria:

1. information about an earlier sudden hearing loss
2. information on chronic middle ear inflammation
3. information on ear surgery (except placement of ventilation tubes in the eardrum)
4. information on dizziness associated with hearing loss and noise
5. information on insomnia
6. current use of oral corticosteroids
7. bilaterally found air-bone gap greater than 15 dB

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: An employer finds workers who meet points 1-5 of study inclusion criteria. A head of the research checks their medical history and includes them in the study if they do not meet any of first six exclusion criteria. A head of the research orally informs these workers at the meeting and helps them to understand and sign a written informed consent for participation in the research. Each of them receive an information about the date of arrival at the place of research and also a unique password that encodes saliva samples, completed questionnaires and electronic and printed findings derived from the assessment of hearing health.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
auditory evoked brainstem response (ABR) characteristics | 1 day
  auditory evoked brainstem response after noise exposure
salivary cortisone concentration | 1 day
  salivary cortisone concentration after noise exposure

CONTACTS AND LOCATIONS:
Overall Officials: Mihael Ries, MD, PhD, Study Director — Department of Otorhinolaryngology and Head and Neck Surgery
Locations (1):
- University Hospital Center Sestre milosrdnice, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No